CLINICAL TRIAL: NCT05996796
Title: Cervical Cancer Screening Based on First-void Urine Self-sampling to Reach un(Der)-Screened Women: Dry Run of the ScreenUrSelf Trial
Brief Title: Dry Run of the ScreenUrSelf Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Antwerp University Hospital (UZA) (Unknown); Centre for Cancer Detection (CvKO) (Unknown); Sciensano (Other Government)
Responsible Party: Principal Investigator, Pierre Van Damme, Principal Investigator, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B3002023000038
Record Dates: First submitted 2023-08-02; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia; Human Papilloma Virus; HPV-Related Cervical Carcinoma
Keywords: Biomarker; First-void urine; Vaginal sample; Screening; Triage; Self-sampling
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Opt-out first-void urine (Experimental): Women will receive a first-void urine self-sampling study package at home.
  The study package will include an invitation letter/informed consent form, information brochure, first-void urine self-sampling device, safety bag with absorbent paper, pre-stamped return envelope, and instructions explaining how to collect the sample and send it to the lab.
  Interventions: Device: Colli-Pee Small Volumes
- Opt-in first-void urine (Experimental): Women will receive a letter at home with instructions how to order (via phone, e-mail, or webform) a first-void urine self-sampling study package.
  The study package will include an invitation letter/informed consent form, information brochure, first-void urine self-sampling device, safety bag with absorbent paper, pre-stamped return envelope, and instructions explaining how to collect the sample and send it to the lab.
  Interventions: Device: Colli-Pee Small Volumes
- Opt-out vaginal self-sample (Experimental): Women will receive a vaginal self-sampling study package at home.
  The study package will include an invitation letter/informed consent form, information brochure, vaginal self-sampling device, safety bag with absorbent paper, pre-stamped return envelope, and instructions explaining how to collect the sample and send it to the lab.
  Interventions: Device: Evalyn Brush
- Opt-in vaginal self-sample (Experimental): Women will receive a letter at home with instructions how to order (via phone, e-mail, or webform) a vaginal self-sampling study package.
  The study package will include an invitation letter/informed consent form, information brochure, vaginal self-sampling device, safety bag with absorbent paper, pre-stamped return envelope, and instructions explaining how to collect the sample and send it to the lab.
  Interventions: Device: Evalyn Brush

INTERVENTIONS:
Device: Colli-Pee Small Volumes — Women will self-collect a first-void urine sample at home upon receipt of the study package using the Colli-Pee Small Volumes (10 mL) device (Novosanis, Belgium). The collector tube is prefilled with a preservative (UCM, Novosanis, Belgium). Women will send the collector vial containing first-void urine along with the informed consent form to the laboratory at University of Antwerp using the prestamped envelope.
  Arms: Opt-in first-void urine; Opt-out first-void urine
Device: Evalyn Brush — Women will self-collect a vaginal sample at home upon receipt of the study package using the Evalyn Brush device (Rovers Medical Devices, The Netherlands). Women will send the used brush along with the informed consent form to the laboratory at University of Antwerp using the prestamped envelope.
  Arms: Opt-in vaginal self-sample; Opt-out vaginal self-sample

SUMMARY:
The proposed study is the Dry Run preceding the ScreenUrSelf trial.

DETAILED DESCRIPTION:
The ScreenUrSelf trial will be embedded in the Flemish organized cervical cancer screening program. The goal of ScreenUrSelf is to reach women who are eligible but do not participate in cervical cancer screening, by offering two self-sampling methods (first-void urine and vaginal) in an opt-in and -out strategy (total of four interventions) to collect samples for primary high-risk (hr) Human Papillomavirus (HPV) testing, and if positive, reflex 1) cytology on a Pap smear (standard of care) and 2) methylation marker triage (index test). The two control arms include 1) no intervention; and 2) sending (recall) invitation letters to women, inviting them to make an appointment for a Pap smear (i.e., current practice within the organized cervical cancer screening program in Flanders).

The Dry Run which is the subject of this clinical trial will test the study materials and data flows developed for the interventional study arms (C, D, E and F) of the ScreenUrSelf trial. The primary outcome of the Dry Run is to check if the flow for data- and sample collection is ready for start of the ScreenUrSelf trial, and if optimizations are deemed necessary before start of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for cervical cancer screening within the organized Population-based Screening Program in Flanders:

  * Female
  * Residing in Flanders, Belgium
  * No history of total hysterectomy
  * No (former) diagnosis of cervical or uterine cancer
  * 30 - 64 years old (birth year 1959 - 1992)

Exclusion Criteria:

* Being pregnant or 6 weeks postpartum (self-reported after receiving the study letter/package)
* Participation during menstruation or within the 3 following days is a contraindication
* Not able to understand the study materials and participation form (informed consent form)

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
HPV DNA using the Riatol qPCR HPV genotyping assay | Through study completion, an average of 1 year
  HPV DNA concentration [copies/µl DNA] in self-samples from all study participants.

SECONDARY OUTCOMES:
Human DNA (Beta-globin) using the Riatol qPCR HPV genotyping assay | Through study completion, an average of 1 year
  Human DNA concentration [copies/µl DNA] in self-samples from all study participants
Preferences | Through study completion, an average of 1 year
  Preferences and attitudes of women regarding self-sampling (measured using a questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Universiteit Antwerpen, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No